CLINICAL TRIAL: NCT02513771
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial of a Dipeptidyl Peptidase-4 Inhibitor (Sitagliptin, Januvia) for Reducing Inflammation and Immune Activation in HIV-Infected Men and Women: A Multicenter Trial of the AIDS Clinical Trials Group (ACTG)
Brief Title: Sitagliptin for Reducing Inflammation and Immune Activation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5346; UM1AI068636 (NIH)
Record Dates: First submitted 2015-07-13; First posted 2015-08-03 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: HIV-1 Infection
Keywords: Sitagliptin; Inflammation; Immune activation; Viral suppression; HIV-1; Immunology biomarkers; sCD14
MeSH Terms: conditions — Inflammation | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin Arm (Active Comparator): Sitagliptin (Januvia) 100 mg one tablet daily p.o. for 16 weeks, followed by a 4-week post-treatment follow-up.
  Interventions: Drug: Sitagliptin
- Placebo Arm (Placebo Comparator): Placebo for sitagliptin one tablet daily p.o.for 16 weeks, followed by a 4-week post-treatment follow-up.
  Interventions: Drug: Placebo for sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 100 mg one tablet taken orally daily for 16 weeks, followed by a 4-week post-treatment follow-up
  Other Names: Januvia
  Arms: Sitagliptin Arm
Drug: Placebo for sitagliptin — One tablet taken orally daily for 16 weeks, followed by a 4-week post-treatment follow-up.
  Other Names: Placebo
  Arms: Placebo Arm

SUMMARY:
The purpose of the study is to evaluate whether sitagliptin (Januvia is the brand name for sitagliptin) reduces inflammation and immune activation markers in HIV-infected men and women when compared to a placebo (inactive medication like a dummy pill). The study evaluated whether taking 100 mg of sitagliptin by mouth daily for 16 weeks is safe and effective for HIV-infected persons on antiretroviral therapy (ART) who do not have diabetes. Sitagliptin is a medication that is used to treat people with diabetes (high blood sugar) but also may reduce inflammation in the body.

DETAILED DESCRIPTION:
ACTG A5346 is a phase II, randomized, double-blinded, placebo-controlled, trial of sitagliptin 100 mg vs. placebo for 16 weeks followed by a 4-week post-intervention follow-up. A5346 studied whether sitagliptin reduced plasma concentrations of sCD14 in HIV-infected men and women ≥18 years of age who were on suppressive ART with HIV-1 RNA below the limit of quantification at screening and for at least the prior 48 weeks. Participants were randomized 1:1 to Sitagliptin arm vs. Placebo arm, and were stratified by screening CD4 count (100-350 vs. >350 cells/mm^3) and statin use (on statins vs. not on statins).

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection.
* Currently on an antiretroviral regimen consisting of at least 2 NRTIs and either a protease inhibitor boosted with low dose ritonavir, an integrase inhibitor, or an NNRTI. (Other ART regimens may be acceptable. Sites must consult the protocol team for approval)
* Currently on continuous ART for ≥48 weeks prior to study entry with no interruption longer than 7 consecutive days during that period.
* Plasma HIV-1 RNA levels below 75 copies/mL for at least 48 weeks prior to study entry. The participant must have a minimum of two values in the last 48 weeks obtained >30 days apart, with the most recent value obtained within 90 days prior to entry. (Single determinations that are between the assay quantification limit and 500 copies/mL (i.e., "blips") are allowed as long as the preceding and subsequent determinations are below the level of quantification).
* CD4+ cell count ≥100 cells/mm^3 obtained within 90 days prior to study entry.
* The following laboratory values obtained within 90 days prior to entry.

  * Absolute neutrophil count (ANC) ≥750/mm^3
  * Hemoglobin ≥8.0 g/dL
  * Platelet count ≥50,000/mm^3
  * Calculated creatinine clearance (CrCl) ≥60 mL/min as estimated by the Cockroft-Gault formula NOTE: Calculation for the Cockcroft-Gault equation is available at https://www.fstrf.org/apps/cfmx/apps/common/Portal/index.cfm
  * Aspartate aminotransferase (AST) (SGOT) ≤5 x upper limit of normal (ULN).
  * alanine aminotransferase (ALT) (SGPT) ≤5 x ULN.
  * alkaline phosphatase ≤5 x ULN.
  * Total bilirubin ≤2.5 x ULN (if the participant is receiving atazanavir, a total bilirubin of ≤5 x ULN is acceptable).
  * Hemoglobin A1C ≤6.5%
* For females of reproductive potential, adequate contraception.
* Karnofsky performance score ≥70 within 90 days prior to entry.
* Ability and willingness of participant or legal guardian/representative to provide informed consent.
* Participants on statin therapy must be stable on the same dose for at least the prior 12 weeks with no anticipated change in statin or dose during the intervention.

Exclusion Criteria:

* Change in the ART regimen within the 12 weeks prior to study entry, or anticipated/intended modification of ART during the study period.
* Two or more HIV-1 RNA determinations >200 copies/mL within the 48 week period prior to study entry.
* History of clinical pancreatitis or diabetes mellitus diagnosed by a medical provider.
* Acute or chronic liver disease with evidence of cirrhosis or portal hypertension.
* Chronic hepatitis C (defined as HCV antibody positive and HCV RNA detectable).
* History of chronic hepatitis B (defined as surface antibody negative, surface antigen positive, and/or HBV DNA detectable).
* Use of any immunomodulator, HIV vaccine, investigational therapy, or anti-TNF therapies within 90 days prior to study entry.
* Active malignancy with expected need for systemic chemotherapy or radiation therapy during the study period.
* Use of human growth hormone, tesamorelin, testosterone or anabolic steroids within 90 days prior to study entry (except chronic, stable, replacement dosages in men with diagnosed hypogonadism is allowed).
* Pregnant or breastfeeding.
* Use of any anti-diabetic medication or GLP-1 analogues within the 12 weeks prior to study entry.
* Current diagnosis of congestive heart failure.
* Known allergy/sensitivity or any hypersensitivity to components of the study drug or its formulation.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 90 days prior to entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12-13 (Actual); Study Completion 2017-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dube, MD, Study Chair — University of Southern California; Kevin Yarasheski, PhD, Study Chair — Washington University School of Medicine
Locations (16):
- United States (16):
  - University of Southern California (1201), Los Angeles, California
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - Whitman Walker Health CRS (31791), Washington D.C., District of Columbia
  - Washington University CRS (2101), St Louis, Missouri
  - Cornell CRS (7804), New York, New York
  - Columbia Physicians and Surgeons CRS (30329), New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (31787), Rochester, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Greensboro CRS (3203), Greensboro, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pittsburgh CRS (1001), Pittsburgh, Pennsylvania
  - Houston AIDS Research Team CRS (31473), Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant was enrolled on October 20, 2015. Accrual to the study closed on August 24, 2016, with 15 U.S sites registered and enrolled participants.
Pre-assignment Details: Participants were randomized 1:1 to Sitagliptin and Placebo arms. Randomization was stratified by screening CD4 (100-350 vs >350 cells/mm^3) and statin use.
Period: Overall Study
Arm/Group | Sitagliptin Arm | Placebo Arm
Started | 45 | 45
Completed | 43 | 44
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Not being able to get to clinic | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin Arm | Placebo Arm | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [40 to 56] | 50 [45 to 55] | 51 [44 to 56]
Age, Customized [Count of Participants; unit: Participants]
  18-39 years | 11 | 6 | 17
  40-59 years | 27 | 32 | 59
  >=60 years | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 38 | 36 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 23 | 18 | 41
  Non-Hispanic Black | 15 | 19 | 34
  Hispanic (Regardless of Race) | 7 | 7 | 14
  more than one race | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 45 | 90
IV drug use [Count of Participants; unit: Participants]
  Never | 44 | 42 | 86
  Previously | 1 | 3 | 4
CD4 count [Median (Inter-Quartile Range); unit: cells/mm^3] — CD4 count at entry Population: Enrolled participants with available baseline CD4 count. One participant had missing CD4 count at baseline due to missing blood samples.
  cells/mm^3
    number analyzed (Participants) | 45 | 44 | 89
    (all) | 609 [323 to 796] | 551 [313 to 801] | 586 [317 to 796]
Baseline sCD14 [Median (Inter-Quartile Range); unit: log10 pg/mL] — sCD14 is the primary endpoint of the study. Baseline sCD14 is the average of pre-entry and entry values Population: As-treated population limited to participants who had baseline and week 15 measurements, completed study treatment with no more than 34 cumulative days of treatment interruption, did not use prohibited medications, did not have a confirmed virologic failure at or prior to week 16 (see protocol 6.2.3).
  log10 pg/mL
    number analyzed (Participants) | 42 | 42 | 84
    (all) | 6.39 [6.31 to 6.44] | 6.38 [6.33 to 6.48] | 6.39 [6.32 to 6.46]

OUTCOME MEASURES:

1. Primary Outcome: Change in sCD14 From Baseline to Week 15/16
Description: sCD14 (soluble cluster of differentiation 14) is a biomarker of gut microbial translocation and monocyte/macrophage activation.
  The outcome measures are changes in log10 transformed sCD14 from baseline to week 15/16 (week 15/16 - baseline) Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 15 and week 16 were averaged for week 15/16.
Time Frame: Pre-entry, Week 0, Week 15, Week 16
Population: As-treated population limited to participants who had baseline and week 15/16 measurements, completed study treatment with no more than 34 cumulative days of treatment interruption, did not use prohibited medications, did not have a confirmed virologic failure at or prior to week 16 (see protocol 6.2.3).
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 42
log10 pg/mL | -0.03 [-0.06 to 0.02] | -0.03 [-0.08 to 0.02]
Statistical Analysis 1: Comparison: Sitagliptin Arm vs Placebo Arm; Null hypothesis: There is no difference between the two arms in the change in sCD14 from baseline to week 15/16; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney); Stratified Wilcoxon rank-sum test stratified by screening CD4 count (<= or > 350 cells/mm^3) and statin use

2. Secondary Outcome: Change in sCD14 From Week 15/16 to Week 20
Description: sCD14 (soluble cluster of differentiation 14) is a biomarker of gut microbial translocation and monocyte/macrophage activation.
  The outcome measures are changes in log10 transformed sCD14 from week 15/16 to week 20 (week 20 - week 15/16).
  Levels measured at week 15 and week 16 were averaged for week 15/16.
Time Frame: Week 15, week 16, week 20
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 42
log10 pg/mL | 0.04 [-0.02 to 0.13] | 0.02 [-0.10 to 0.11]

3. Secondary Outcome: Change in sCD163
Description: sCD163 (soluble CD 163) is a marker of macrophage activation and arterial inflammation.
  Change in log10 transformed sCD163 from Week 0 to week 15 (week 15 - week 0), and from week 15 to week 20 (week 20 - week 15).
Time Frame: Week 0, week 15, week 20
Population: As-treated population limited to participants who had baseline and week 15 measurements, completed study treatment with no more than 34 cumulative days of treatment interruption, did not use prohibited medications, did not have a confirmed virologic failure at or prior to week 16 (see protocol 6.2.3).
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 42
log10 ng/mL
  Change from week 0 to week 15 | -0.03 [-0.06 to 0.02] | -0.02 [-0.09 to 0.03]
  Change from week 15 to week 20 | 0.01 [-0.02 to 0.05] | 0.00 [-0.06 to 0.05]

4. Secondary Outcome: Change in sCD26
Description: sCD26 (soluble cluster of differentiation 26) is an enzyme that metabolizes DPP-4 (dipeptidyl peptidase-4), an enzyme that is inhibited by sitagliptin.
  Change in log10 transformed sCD26 from Week 0 to week 15 (week 15 - week 0), and from week 15 to week 20 (week 20 - week 15).
Time Frame: Week 0, week 15, week 20
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 42
log10 ng/mL
  Change from week 0 to week 15 | -0.16 [-0.37 to 0.07] | -0.16 [-0.52 to 0.09]
  Change from week 15 to week 20 | 0.08 [-0.28 to 0.24] | 0.04 [-0.16 to 0.26]

5. Secondary Outcome: Change in IL-6
Description: IL-6 (Interleukin-6) is a biomarker of systemic inflammation. Change in log10 transformed IL-6 from Week 0 to week 15 (week 15 - week 0), and from week 15 to week 20 (week 20 - week 15).
Time Frame: Week 0, week 15, week 20
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 42
log10 pg/mL
  Change from week 0 to week 15 | 0.00 [-0.12 to 0.11] | 0.00 [-0.11 to 0.14]
  Change from week 15 to week 20 | -0.06 [-0.11 to 0.08] | 0.01 [-0.10 to 0.12]

6. Secondary Outcome: Change in hsCRP
Description: hsCRP (high-sensitivity C-reactive protein) is a biomarker of inflammation. Change in log10 transformed hsCRP from Week 0 to week 15 (week 15 - week 0), and from week 15 to week 20 (week 20 - week 15).
Time Frame: Week 0, week 15, week 20
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 42
log10 ng/mL
  Change from week 0 to week 15 | -0.08 [-0.18 to 0.06] | -0.05 [-0.22 to 0.10]
  Change from week 15 to week 20 | -0.02 [-0.22 to 0.09] | -0.01 [-0.19 to 0.18]

7. Secondary Outcome: Change in sTNF-r1
Description: sTNF-r1 (soluble tumour necrosis alpha receptor 1) is a biomarker of inflammation.
  Change in log10 transformed sTNF-r1 from Week 0 to week 15 (week 15 - week 0), and from week 15 to week 20 (week 20 - week 15).
Time Frame: Week 0, week 15, week 20
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 42
log10 pg/mL
  Change from week 0 to week 15 | -0.01 [-0.05 to 0.04] | -0.04 [-0.06 to 0.00]
  Change from week 15 to week 20 | 0.00 [-0.03 to 0.06] | -0.01 [-0.05 to 0.09]

8. Secondary Outcome: Change in sTNF-r2
Description: sTNF-r2 (soluble tumour necrosis alpha receptor 2) is a biomarker of inflammation.
  Change in log10 transformed sTNF-r2 from Week 0 to week 15 (week 15 - week 0), and from week 15 to week 20 (week 20 - week 15).
Time Frame: Week 0, week 15, week 20
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 42
log10 pg/mL
  Change from week 0 to week 15 | -0.05 [-0.14 to 0.13] | -0.06 [-0.13 to 0.04]
  Change from week 15 to week 20 | 0.06 [-0.08 to 0.20] | 0.05 [-0.07 to 0.21]

9. Secondary Outcome: Change in IP-10
Description: IP-10 (also known as CXCL10) is a biomarker implicated in cardiovascular disease.
  Change in log10 transformed IP-10 from Week 0 to week 15 (week 15 - week 0), and from week 15 to week 20 (week 20 - week 15).
Time Frame: Week 0, week 15, week 20
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 42
log10 pg/mL
  Change from week 0 to week 15 | -0.31 [-0.40 to -0.15] | -0.01 [-0.09 to 0.12]
  Change from week 15 to week 20 | 0.23 [0.17 to 0.40] | 0.02 [-0.09 to 0.08]

10. Secondary Outcome: Change in CD4+/CD8+ T-cell Ratio
Description: CD4+/CD8+ T-cell ratio change from week 0 to week 15 (week 15 - week 0). Note that CD4 and CD8 were not evaluated at week 20 in this study.
Time Frame: Week 0 and week 15
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 42
ratio | 0.00 [-0.11 to 0.04] | 0.02 [-0.04 to 0.08]

11. Secondary Outcome: Change in CD4+ T-cell Activation
Description: Level of CD4+ T-cell activation was determined by measuring the percentage of cells that expressed both the activation marker CD38+ and Human leukocyte antigen (HLA)-DR+.
  The endpoint is measuring the change from week 0 to week 15 (week 15 - week 0) and change from week 15 to week 20 (week 20 - week 15).
  Data for cellular markers are not available as of December 2017. These data are based on immunology assays which were tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 1 month after the primary complete date. Please note that these secondary outcomes were not included in the primary analyses. There are many outcomes in this study and the immunology lab had to give priority to the assays planned to be included in the primary manuscript. Results will be entered once the data is complete and analyzed.
Time Frame: Week 0, week 15, week 20
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 40
percentage of cells
  change from baseline to week 15: number analyzed (Participants) | 41 | 40
  change from baseline to week 15 | 0.12 [-0.15 to 0.52] | 0.08 [-0.41 to 0.43]
  change from week 15 to week 20 | 0.07 [-0.28 to 0.60] | 0.06 [-0.47 to 0.38]

12. Secondary Outcome: Change in CD8+ T-cell Activation
Description: Level of CD8+ T-cell activation was determined by measuring the percentage of cells that expressed both the activation marker CD38+ and Human leukocyte antigen (HLA)-DR+.
  The endpoint is measuring the change from week 0 to week 15 (week 15 - week 0) and change from week 15 to week 20 (week 20 - week 15).
  Data for cellular markers are not available as of December 2017. These data are based on immunology assays which were tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 1 month after the primary complete date. Please note that these secondary outcomes were not included in the primary analyses. There are many outcomes in this study and the immunology lab had to give priority to the assays planned to be included in the primary manuscript. Results will be entered once the data is complete and analyzed.
Time Frame: Week 0, week 15, week 20
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 40
percentage of cells
  change from baseline to week 15: number analyzed (Participants) | 41 | 40
  change from baseline to week 15 | 0.03 [-0.90 to 1.83] | -0.27 [-1.11 to 1.33]
  change from week 15 to week 20 | 0.11 [-0.70 to 1.90] | -0.29 [-1.12 to 1.17]

13. Secondary Outcome: Change in %CD14+/CD16- (Classical Monocytes)
Description: CD14+/CD16- is the percentage of cells that expressed CD14 and low CD16 in total monocytes (also known as classical monocytes).
  This endpoint is measuring the change from week 0 to week 15 (week 15 - week 0) and change from week 15 to week 20 (week 20 - week 15).
  Data for cellular markers are not available as of November 2017. The study team prioritized completion of the soluble markers (including the primary outcome measure), which are reported herein, over the completion of the cellular markers. Results will be entered once the data is complete and analyzed.
Time Frame: Week 0, week 15, week 20
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 40
percentage of cells
  change from baseline to week 15: number analyzed (Participants) | 41 | 40
  change from baseline to week 15 | -2.30 [-6.20 to 3.20] | -0.80 [-4.75 to 2.75]
  change from week 15 to week 20 | 0.40 [-2.40 to 6.10] | -1.00 [-4.50 to 4.95]

14. Secondary Outcome: Change in %CD14+/CD16+ (Intermediate Monocytes)
Description: %CD14+/CD16+ is the percentage of cells that expressed both CD14 and CD16 in total monocytes (also known as intermediate monocytes).
  This endpoint is measuring the change from week 0 to week 15 (week 15 - week 0) and change from week 15 to week 20 (week 20 - week 15).
  Data for cellular markers are not available as of December 2017. These data are based on immunology assays which were tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 1 month after the primary complete date. Please note that these secondary outcomes were not included in the primary analyses. There are many outcomes in this study and the immunology lab had to give priority to the assays planned to be included in the primary manuscript. Results will be entered once the data is complete and analyzed.
Time Frame: Week 0, week 15, week 20
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 40
percentage of cells
  change from baseline to week 15: number analyzed (Participants) | 41 | 40
  change from baseline to week 15 | 0.87 [-1.32 to 3.08] | -0.12 [-2.33 to 1.97]
  change from week 15 to week 20 | -0.65 [-2.86 to 0.98] | -0.19 [-1.50 to 1.37]

15. Secondary Outcome: Change in %CD14dim/CD16++ (Non-classical Monocytes)
Description: %CD14dim/CD16++ is the percentage of cells that expressed low levels of CD14dim and high levels of CD16++ in total monocytes (also known as non-classical monocytes).
  This endpoint is measuring the change from week 0 to week 15 (week 15 - week 0) and change from week 15 to week 20 (week 20 - week 15).
  Data for cellular markers are not available as of December 2017. These data are based on immunology assays which were tested in batch to minimize variability. Due to batch testing, shipment of samples for testing could not begin until after the study follow-up completion, which was 1 month after the primary complete date. Please note that these secondary outcomes were not included in the primary analyses. There are many outcomes in this study and the immunology lab had to give priority to the assays planned to be included in the primary manuscript. Results will be entered once the data is complete and analyzed.
Time Frame: Week 0, week 15, week 20
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 42 | 40
percentage of cells
  change from baseline to week 15: number analyzed (Participants) | 41 | 40
  change from baseline to week 15 | 0.31 [-1.02 to 2.05] | -0.03 [-2.08 to 2.31]
  change from week 15 to week 20 | -0.37 [-1.95 to 1.76] | 0.12 [-1.16 to 2.89]

16. Secondary Outcome: Number of Participants With Grade ≥2 Adverse Events Related to Study Drug
Description: The DAIDS Adverse Event Grading Table, Version 2.0, was used for grading of AEs
Time Frame: From study entry to end of study (Week 20)
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 45 | 45
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) reported from first dose of study treatment until study completion at 20 weeks
Description: Expedited adverse event (EAE) reporting followed the Division of AIDS (DAIDS) EAE Manual under the SAE Reporting Category and including fetal losses. Events were graded (1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death) according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Clarification Aug 2009.
Groups:
- Sitagliptin: Sitagliptin (Januvia) 100 mg one tablet daily p.o. for 16 weeks, followed by a 4-week post-treatment follow-up.
- Placebo: Placebo for sitagliptin one tablet daily p.o.for 16 weeks, followed by a 4-week post-treatment follow-up.
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/45 | 2/45
Other Adverse Events (participants affected / at risk) | 20/45 | 24/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=45) | Placebo (N=45)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=45) | Placebo (N=45)
Nausea (Gastrointestinal disorders) | 1 | 3
Fatigue (General disorders) | 1 | 3
Pyrexia (General disorders) | 1 | 3
Alanine aminotransferase (Investigations) | 5 | 2
Aspartate aminotransferase (Investigations) | 3 | 3
Blood bilirubin increased (Investigations) | 3 | 3
Blood creatinine abnormal (Investigations) | 4 | 5
Blood glucose decreased (Investigations) | 3 | 1
Blood glucose increased (Investigations) | 1 | 4
Blood uric acid increased (Investigations) | 1 | 3
Haemoglobin decreased (Investigations) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.